CLINICAL TRIAL: NCT00226538
Title: Prediction of Potential Drug Interaction With CYP2C9 Substrate by Using Phenytoin Metabolic Ratio as a Marker of Its Activity in-Vivo.
Brief Title: Prediction of Drug Interactions With CYP2C9 Substrates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: yc19555-HMO-CTIL
Record Dates: First submitted 2005-09-12; First posted 2005-09-27 (Estimated); Last update posted 2008-10-29 (Estimated); Status verified 2008-10

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — Phenytoin; Rifampin; Diclofenac; Fluconazole

INTERVENTIONS:
Drug: Phenytoin
Drug: Rifampicin
Drug: Diclophenac
Drug: Fluconazole

SUMMARY:
CYP2C9, is one of the major drug metabolism enzymes accounting for about 20% of the hepatic cytochrome P450 content and being second only to CYP3A4.

The proposed study will explore different possible drug interactions with CYP2C9 substrates by evaluating the effect of prototype inducers and inhibitors on the phenotypic trait measurement. It is expected that the identification of drugs that might interact with CYP2C9 substrates will be used to rationalize future drug interaction studies designed to evaluate the actual magnitude of effect and its clinical implications. This approach should be particularly useful when applied to those CYP2C9 drugs characterized by a narrow therapeutic index (i.e. warfarin).

This study will consist of three study periods separated from each other by a two weeks washout period. In the course of the study the subjects will receive in a double blind, crossover fashion, rifampin 300 mg. twice daily, diclofenac 50 mg twice daily. and fluconazole 200 mg. twice daily, each for one week. All drugs will be administered as identical looking tablets that will be prepared at the pharmacy of the Hadassah University Hospital and their order of administration will be randomized.On the day prior to, on day 6 of and 7 days following each drug period, the activity of CYP2C9 will be evaluated by the administration of a single phenytoin 300 mg. dose. The subjects will be requested to collect their urine for 24 hours and a single blood sample will be obtained 12 hours post phenytoin intake.

ELIGIBILITY:
Inclusion Criteria:

* Age range 20-50
* Absence of significant disease states

Exclusion Criteria:

* Known hypersensitivity to one of the drugs used in the study
* Significant disease states
* Regular use of drugs (including birth control pills)

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 1999-08

PRIMARY OUTCOMES:
Phenytoin metabolic ratio prior to and following exposure to fluconazole, diclophenac and rifampicin.

CONTACTS AND LOCATIONS:
Overall Officials: Yoseph Caraco, MD, Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel